CLINICAL TRIAL: NCT06186791
Title: Self-directed Dying in the Netherlands by Voluntarily Stopping Eating and Drinking or Independently Intake of Lethal Medication Attended by a Confidant.
Brief Title: Self-directed Dying in the Netherlands
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Agnes van der Heide, Prof. dr., Erasmus Medical Center
Other Study IDs: 10894
Record Dates: First submitted 2023-10-23; First posted 2024-01-02 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-12

CONDITIONS: Suicide, Assisted; Fasting; Decision Making
Keywords: Wish to hasten death; Voluntary stopping eating and drinking; Independently intake of lethal medication (attended by a confident); Self determination; Personal autonomy
MeSH Terms: conditions — Suicide, Assisted; Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In 2007, the frequency of so-called 'self-directed dying' in the Netherlands was investigated, that is, the voluntary cessation of eating and drinking or the taking of lethal self-collected medication. This research has not been repeated yet. Since 2007 there have been major developments regarding assisted and non-assisted dying, including the issue of a guideline by the KNMG and the endorsement by various political parties of a proposal for a new law on assistance in dying. There has also been much societal debate on euthanasia and assisted suicide as regulated by the Termination of Life on Request and Assisted Suicide (Review Procedures) Act. These developments may have had an influence on the frequency of self-directed dying.

The primary objective of this cross-sectional questionnaire study with add-on qualitative interviews is to estimate how many people die each year in the Netherlands by either voluntarily stopping eating or drinking (VSED) or intentional intake of lethal medication attended by a confidant (ILMC). Secondary objectives include studying whether this number has changed since 2007; exploring possible explanations for changes in frequencies; and providing insight in the quality of dying of people who choose self-directed dying.

To this end an online questionnaire will be sent out to a randomly drawn sample (n ≈ 37 500) from a large representative panel (NIPObase) of the Dutch adult population. A two-stage screening procedure will be used to check whether the experiences of the respondents represent a death VSED or by ILMC. The data will be analysed using quantitative software SPSS. From the respondents who indicate that they are willing to be interviewed, a sample will be taken from each group, 20 from VSED and 20 from ILMC. Interviews will be conducted by an experienced interviewer. The interviews are focused on better understanding people's choice for a self-directed death and on the perceived quality of the dying process for both methods. The interviews will be audio recorded and thematically analysed using qualitative software (N-Vivo).

DETAILED DESCRIPTION:
The frequency of both types of self-directed deaths in the population can be estimated with the standard weighting method that is used by Statistics Netherlands (CBS) in estimating the annual frequency of relatively rare events such as traffic incidents. The investigators will use an adapted standard weighting. Each informant is weighted by the inverse of 1 (the informant) plus the number of other individuals who had been confided by the deceased person about their intention to hasten death by VSED or ILMC. The estimated number of cases will be computed for the responding part of the sample. For the frequency estimation, the investigators will use the number of informants on a death by VSED or ILMC in the five years from 1 January 2018 to 31 December 2022, because reports about cases before 2018 are considered less reliable. The annual frequency of VSED and ILMC can then be computed as the estimated proportion of reported cases in the sample (i.e. weighted sum of informants on VSED deaths and ILMC deaths respectively divided by sample size corrected for non-response), multiplied by the total number of Dutch adults minus non-western adults (underrepresented in the sample) and divided by the five years covered by the informants. The Poisson distribution will be used in calculating the 95% Confidence Intervals (CIs).

Secondary outcomes will be mainly described in frequency tables, using standard statistical analysis.

The interview transcripts will be analysed thematically using NVivo software.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Be able to speak and read Dutch
* Have given informed consent to participation

Exclusion Criteria:

* Younger than 18 years
* Not able to speak and read Dutch
* Not giving informed consent to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample (n ≈ 37 500) of Dutch adults over the age of 18 will be randomly drawn from a large panel of adults willing to participate in questionnaire research. The panel is representative of the Dutch adult population in terms of gender, age, education and geographical location.
Sampling Method: Probability Sample
Enrollment: 37500 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Frequency of annual self-directed deaths | January 2024 - March 2024
  An estimate of the number of people who die each year by voluntary stopping eating and drinking, and an estimate of the number of people who die each year by independent intake of lethal medication attended by a confidant.

SECONDARY OUTCOMES:
Comparison of estimates of self-directed deaths | May 2024
  A comparison of current estimates with the estimated numbers of self-directed deaths in 2007
Changes in frequencies | May - September 2024
  An exploration of possible explanations for changes in frequencies
Decision-making process and quality of dying | June - September 2024
  Providing insight in the decision-making process and the quality of dying of people who choose self-directed dying.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes van der Heide, prof. dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chabot BE, Goedhart A. A survey of self-directed dying attended by proxies in the Dutch population. Soc Sci Med. 2009 May;68(10):1745-51. doi: 10.1016/j.socscimed.2009.03.005. Epub 2009 Apr 15. PMID 19375206
- [Derived] Bosma F, Stoppelenburg A, van der Heide A, van de Vathorst S. Frequency of self-directed dying in the Netherlands: research protocol of a cross-sectional mixed-methods study. BMJ Open. 2024 Apr 29;14(4):e085240. doi: 10.1136/bmjopen-2024-085240. PMID 38684276